CLINICAL TRIAL: NCT02241746
Title: Malnutrition in Chinese Hospitalized Patients and Optimizing the Usage of Nutritional Screening Tools
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yexuan TAO, associate chief physician, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XHEC-C-2014-088
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- malnutrition
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
The purpose of this study is:

* to diagnose malnutrition in Chinese hospitalized patients with four nutritional screening tools: mini-nutritional assessment - short form, subjective global assessment, malnutrition universal screening tool and nutritional risk screening 2002.
* to optimize the usage of nutritional screening tools based on data-mining methods.

ELIGIBILITY:
Inclusion Criteria:

* Ages≥18; admitted to hospital≥24h and did not receive operation until 8.am next day.

Exclusion Criteria:

* Patients who were pregnant or breast-feeding, and those who could not be interviewed or provide informed consent were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary general hospital
Sampling Method: Non-Probability Sample
Enrollment: 856 (Actual)
Dates: Start 2012-08; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
prevalence of malnutrition on admission detected by the four nutritional screening tools | up to 4 weeks
  The measure of prevalence of malnutrition on admission is a composite outcome measure. In our study, we used four nutritional screening tools: MUST(malnutrition universal screening tool), SGA(subjective global assessment), MNA-SF(mini-nutritional assessment-short form) and NRS2002(nutritional risk screening 2002) to assess the malnutrition risk among Chinese hospitalized patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China